CLINICAL TRIAL: NCT02496247
Title: Effectiveness of Canned Herring for Prevention of Childhood Malnutrition During the Early Rainy Season in Rural Guinea-Bissau
Brief Title: Canned Herring for Prevention of Childhood Malnutrition During the Early Rainy Season in Rural Guinea-Bissau
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Global Food & Nutrition Inc. (Other)
Collaborators: Alaska Seafood Marketing Institute (Unknown); International Partnership for Human Development (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GFN GB 2015
Record Dates: First submitted 2015-04-30; First posted 2015-07-14 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Malnutrition; Undernutrition
Keywords: malnutrition; undernutrition; Z-score; Guinea-Bissau; food aid
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Herring (Experimental): Participants in this arm will receive the Canned Herring intervention. Families with children in this study arm will receive a weekly ration of herring throughout the 8-10 week study period (2 cans herring/day per study child), which will be distributed weekly by community health workers. Families will be instructed to feed the study child half a can of herring per day (without reducing usual home food given to the child), and to not share the remaining herring with individuals who are in the Delayed Herring study arm. When families come to collect their weekly distribution they will be asked to bring in at least 7 empty herring cans in order to receive the next ration, and will answer a question about how often the child eats the herring.
  Interventions: Other: Canned Herring
- Delayed Herring (Control) (No Intervention): Families with children in this study arm will not receive any herring during the 8-10 week period when Immediate Herring families receive a weekly ration of herring. After the 8-10 week (end line) measurements, an equal amount of herring will be distributed to the family.

INTERVENTIONS:
Other: Canned Herring — Families with children in this study arm will receive a weekly ration of herring throughout the 8-10 week study period (2 cans herring/day per study child).
  Arms: Immediate Herring

SUMMARY:
This study will test the effectiveness of a weekly village distribution of canned herring for prevention of malnutrition in children aged 2-5 years old during a food-insecure time of the year in rural villages in Guinea-Bissau. The study will use community health workers to conduct the herring distribution, making this a test that will provide valuable information on what could become a practical food aid supplementation practice. The primary study hypothesis is that distribution of canned herring as a weekly food supplement to families with young children at the beginning of the rainy season will prevent a seasonal decrease in weight-for-age Z-score (primary variable) of children with mild to moderate malnutrition at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Village leaders willing to allow the study to take place in their village
* Village must have community health workers who are willing to do the weekly distribution of herring to enrolled families and are able to keep the necessary records documenting the distribution.
* Children age 2-5 currently living in a selected village
* Parents willing to participate in the study

Exclusion Criteria:

* There are no eligibility exclusions for this study.
* If a child is identified with severe malnutrition at the baseline measurement, the family will be advised to take the child for treatment rather than participate in the study.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in weight-for-age Z-score | baseline, 8-10 weeks

SECONDARY OUTCOMES:
height-for-age Z-score | baseline, 8-10 weeks
mid upper arm circumference (MUAC) measurement | baseline, 8-10 weeks
  measurement of circumference of the mid upper arm
weight | baseline, 8-10 weeks
height | baseline, 8-10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nina Schlossman, Principal Investigator — Global Food & Nutrition Inc.; Adrian Balan, Principal Investigator — International Partnership for Human Development